CLINICAL TRIAL: NCT02389803
Title: Double Blind, Randomized , Placebo Controlled Study to Evaluate the Effect of Nutritional Supplementation on Growth of Short and Lean Adolescents Boys
Brief Title: Evaluating the Effect of Nutritional Supplementation on Growth of Short and Lean Adolescents Boys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rmc067614ctil
Record Dates: First submitted 2015-03-11; First posted 2015-03-17 (Estimated); Last update posted 2022-02-22 (Actual); Status verified 2019-12

CONDITIONS: Growth Problem; Low Weight; Short Stature
MeSH Terms: conditions — Thinness; Dwarfism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional supplementation standardized formula (Experimental): Powder added to water, containing about 25% of recommended Daily Recommended Intake (DRI) for Calories, high protein (25% of calories) and multi vitamin and mineral (25%-100% of DRI for recommended daily allowance (RDA) or adequate intake )
  Interventions: Dietary Supplement: Nutritional supplementation standardized formula
- Placebo comparator (Placebo Comparator): Low caloric formula (Powder added to water), without added vitamins and mineral
  Interventions: Dietary Supplement: Placebo comparator

INTERVENTIONS:
Dietary Supplement: Nutritional supplementation standardized formula — Powder added to water, containing about 25% of recommended DRI for Calories, high protein (25% of calories) and multi vitamin and mineral (25%-100% of DRI for recommended daily allowance (RDA) or adequate intake )
  Arms: Nutritional supplementation standardized formula
Dietary Supplement: Placebo comparator — Low caloric formula (Powder added to water), without added vitamins and minerals
  Arms: Placebo comparator

SUMMARY:
Study design:

Double blind, randomized, placebo controlled study. Participants will be randomly assigned either to the intervention group or the placebo control group. Randomization for the two study groups will be made in a ratio of 1:1.

The primary objective of the study is to assess the effect of 6-12 months treatment with nutritional supplementation standardized formula, in short and lean boys adolescents on weight Standard Deviation Score (SDS) and height SDS The Secondary Objectives of the study are to assess the effect of 6-12 months treatment with nutritional supplementation standardized formula, in short and lean boys adolescents on BMI SDS, growth velocity, time to puberty, quality of life and self-esteem The study will continue for 6 months of intervention versus active placebo, with additional optional 6 months (an extension period), in which participants at both groups, the intervention and the placebo, will be offered to continue their participation in the study with the study supplement. All analyses of the effect's on primary and secondary outcome measurements will take into account the consumption rate of the study formula/placebo

ELIGIBILITY:
Inclusion Criteria:

* Boys aged ≥10years old
* Prepubertal - Tanner stage 1 (gonadarche) (testicular volume<4)
* Height and weight ≤ 10th percentile for age and gender.
* Height-SDS ≥ -2.5 SDS
* BMI-SDS>-3 SDS
* Low proportion between weight and height
* Signing inform consent forms

Exclusion Criteria:

* Diagnosis of Growth Hormone (GH) Deficiency or treatment with GH
* Any known chronic disease or dysmorphic syndrome including: bone diseases, organic brain diseases, neurological disease, past or current malignancy, chronic cardiac, renal or pulmonary problems
* Any known gastrointestinal disease including malabsorption
* Any known organic reason for growth retardation

Ages: 10 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2015-06; Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Weight SDS (standard deviation score) | At 12 months
Height SDS (standard deviation score) | At 12 months
Weight SDS (standard deviation score) | At 6 months
Height SDS (standard deviation score) | At 6 months

SECONDARY OUTCOMES:
BMI SDS (standard deviation score) | At 12 months
BMI SDS (standard deviation score) | At 6 months
Growth velocity | At 12 months
Growth velocity | At 6 months
Quality of life | At 12 months
  Quality of life measured by Quality of Life Questionnaire
Quality of life | At 6 months
  Quality of life measured by Quality of Life Questionnaire
Self-esteem (Self-Esteem Questionnaire) | At 12 months
  Self-esteem measured by Self-Esteem Questionnaire
Self-esteem (Self-Esteem Questionnaire) | At 6 months
  Self-esteem measured by Self-Esteem Questionnaire

OTHER OUTCOMES:
Time to puberty initiation (Duration of time until testicular volume is at tanner stage >=2) | At 12 months
  Duration of time until testicular volume is at tanner stage >=2
Sleep assessment Questionnaire | At 12 Months
Sleep assessment Questionnaire | At 6 Months
Physical Activity Questionnaire | At 12 months
Study Participation Questionnaire | At 6 months
Study Participation Questionnaire | At 12 months
Family Eating and Activity Habits Questionnaire | At 6 months
Family Eating and Activity Habits Questionnaire | At 12 months
Parents Stands Towards Healthy Lifestyle Questionnaire | At 6 months
Parents Stands Towards Healthy Lifestyle Questionnaire | At 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, Principal Investigator — Schneider Children's Medical Center
Locations (3):
- Israel (3):
  - Soroka Medical Center, Beersheba
  - Schneider Medical Center, Petah Tikva
  - Assaf Harofe Medical Center, Rishon LeZiyyon